CLINICAL TRIAL: NCT00799201
Title: A Prospective, Randomized Trial of Enteral Naloxone Versus a Traditional Bowel Regimen in Prevention of Constipation and Decreased Gastric Motility in Critically Ill Trauma Patients
Brief Title: Enteral Naloxone Versus a Traditional Bowel Regimen for the Prevention of Opioid Induced Constipation in Trauma Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Naloxone became unavailable due to manufacturing shortatges requiring the study to be terminated.
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Audis Bethea, Pharm.D., Clinical Pharmacy Specialist, Trauma/Surgery, CAMC Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07-01-1897
Record Dates: First submitted 2008-11-24; First posted 2008-11-27 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Constipation; Analgesia
Keywords: Enteral nutrition; Constipation; Gastrointestinal motility; Naloxone; Docusate; Bowel stimulant; Stool softener
MeSH Terms: conditions — Constipation; Agnosia | interventions — Naloxone; Dioctyl Sulfosuccinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Control (Experimental): Sennosides liquid 5mL (8.8mg) every 6 hours plus docusate sodium liquid 10mL (100mg) every 12 hours
  Interventions: Drug: Naloxone and Docusate

INTERVENTIONS:
Drug: Naloxone and Docusate — Naloxone 6mg (15 mL) every 6 hours plus docusate sodium liquid 10 mL (100mg) every 12 hours
  Other Names: Narcan; Colace

SUMMARY:
The purpose of this study is to determine if enteral naloxone is more effective than a traditional bowel regimen in the prevention and treatment of constipation and impaired gastric motility in critically ill trauma patients.

DETAILED DESCRIPTION:
Impaired gastric motility and constipation are common issues among patients in the intensive care setting. Contributing factors include trauma, multiple surgical procedures, lack of ambulation, and the use of opiate analgesics to control pain. Common treatments for altered gastric motility and constipation include administration of pro-motility agents, stool softeners and bowel stimulants.

Enteral feeding is considered the safest and most effective way to provide nutrition to critically ill patients. Nutrition can be delayed and/or held when impaired gastric motility and constipation are present. Studies suggest that delays in the administration of nutrition can lead to prolonged ventilator time and increased length of stay in the intensive care setting as well as an increase in mortality.

Naloxone, a competitive opioid antagonist, is most commonly administered systemically to counteract the central and peripheral effects of opioids. When administered enterally naloxone has also been found to increase gastric emptying. Studies in patients receiving enteral feeds with multiple risk factors for altered gastric motility and constipation suggest that administration of enteral naloxone can reduce the incidence and extent of altered gastric motility and aid in defecation while not totally reversing the systemic effects of the opiate being administered. Due to these findings, it appears that enterally administered naloxone would provide a significant advantage over traditional gastrointestinal stimulants in preventing constipation in critically ill patients receiving continuous administration of opiate analgesics. In addition, the use of an enterally administered opiate antagonist may also alleviate the need for routine administration of pro-kinetic agents in order to promote adequate gastrointestinal motility and toleration of enterally administered nutrition. As a result, the comparison of enteral naloxone plus a stool softener versus a traditional bowel regimen containing a stimulant and stool softener will aid in assessing the effectiveness of opiate reversal locally in the gastrointestinal tract in prevention of decreased gastric motility and constipation.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females > 18 years of age and < 65 years of age
* MSICU admission to the trauma service at the General Hospital
* Scheduled for continuous infusion/administration of opiate analgesics for at least 24 hours
* Access for enteral administration of medications and tube feeds
* Initiation of tube feeds

Exclusion Criteria:

* NPO
* Pregnancy
* < 18 years of age or > 65 years of age
* Pancreatitis
* Ileus
* Large bowel obstruction present on plain X-ray or CT scan
* Recent intestinal anastomosis (within 2 weeks)
* Section of large bowel removed (within 2 weeks)
* Contraindications to metaclopramide (Reglan) such as parkinson's disease, tardive dyskinesia, etc.
* Traumatic brain injury with a glasgow coma score of at least 8
* Use of pharmacologic paralytics or neuromuscular blockade (NMB)
* Non-english speaking patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Number of hours until first bowel movement | While the patient is receiving continuous or scheduled narcotics

SECONDARY OUTCOMES:
Residual volume/toleration of feeds | While the patient is receiving continuous or scheduled doses of narcotics
Average number of bowel movements per day | While the patient is receiving continuous or scheduled narcotics
Escalation of opioid dose due to impaired analgesia | While the patient is receiving study medications

CONTACTS AND LOCATIONS:
Overall Officials: Audis Bethea, PharmD, BCPS, Principal Investigator — CAMC Health System
Locations (1):
- Charleston Area Medical Center, General Hospital, Charleston, West Virginia, United States

REFERENCES:
- [Background] Ely EW, Truman B, Shintani A, Thomason JW, Wheeler AP, Gordon S, Francis J, Speroff T, Gautam S, Margolin R, Sessler CN, Dittus RS, Bernard GR. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA. 2003 Jun 11;289(22):2983-91. doi: 10.1001/jama.289.22.2983. PMID 12799407
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Hawryluck LA, Harvey WR, Lemieux-Charles L, Singer PA. Consensus guidelines on analgesia and sedation in dying intensive care unit patients. BMC Med Ethics. 2002 Aug 12;3:E3. doi: 10.1186/1472-6939-3-3. PMID 12171602
- [Background] Jacobi J, Fraser GL, Coursin DB, Riker RR, Fontaine D, Wittbrodt ET, Chalfin DB, Masica MF, Bjerke HS, Coplin WM, Crippen DW, Fuchs BD, Kelleher RM, Marik PE, Nasraway SA Jr, Murray MJ, Peruzzi WT, Lumb PD; Task Force of the American College of Critical Care Medicine (ACCM) of the Society of Critical Care Medicine (SCCM), American Society of Health-System Pharmacists (ASHP), American College of Chest Physicians. Clinical practice guidelines for the sustained use of sedatives and analgesics in the critically ill adult. Crit Care Med. 2002 Jan;30(1):119-41. doi: 10.1097/00003246-200201000-00020. No abstract available. PMID 11902253
- [Background] Thomas MC, Erstad BL. Safety of enteral naloxone and i.v. neostigmine when used to relieve constipation. Am J Health Syst Pharm. 2003 Jun 15;60(12):1264-7. doi: 10.1093/ajhp/60.12.1264. No abstract available. PMID 12845923
- [Background] Meissner W, Schmidt U, Hartmann M, Kath R, Reinhart K. Oral naloxone reverses opioid-associated constipation. Pain. 2000 Jan;84(1):105-109. doi: 10.1016/S0304-3959(99)00185-2. PMID 10601678
- [Background] Liu M, Wittbrodt E. Low-dose oral naloxone reverses opioid-induced constipation and analgesia. J Pain Symptom Manage. 2002 Jan;23(1):48-53. doi: 10.1016/s0885-3924(01)00369-4. PMID 11779668
- [Background] Mixides G, Liebl MG, Bloom K. Enteral administration of naloxone for treatment of opioid-associated intragastric feeding intolerance. Pharmacotherapy. 2004 Feb;24(2):291-4. doi: 10.1592/phco.24.2.291.33149. PMID 14998227
- [Background] Artinian V, Krayem H, DiGiovine B. Effects of early enteral feeding on the outcome of critically ill mechanically ventilated medical patients. Chest. 2006 Apr;129(4):960-7. doi: 10.1378/chest.129.4.960. PMID 16608945
- [Background] Meissner W, Dohrn B, Reinhart K. Enteral naloxone reduces gastric tube reflux and frequency of pneumonia in critical care patients during opioid analgesia. Crit Care Med. 2003 Mar;31(3):776-80. doi: 10.1097/01.CCM.0000053652.80849.9F. PMID 12626983
- [Background] Mostafa SM, Bhandari S, Ritchie G, Gratton N, Wenstone R. Constipation and its implications in the critically ill patient. Br J Anaesth. 2003 Dec;91(6):815-9. doi: 10.1093/bja/aeg275. PMID 14633751